CLINICAL TRIAL: NCT06088485
Title: Erişkin Kistik Fibrozisli Bireylerde Kemik Mineral Yoğunluğunun Postür, Solunum Fonksiyonları ve Fonksiyonel Egzersiz Kapasitesi Üzerine Etkisi
Brief Title: The Effect of Bone Mineral Density in Patients With Adult Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: GO22/126
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis; Postural Defect; Pulmonary Disease; Physical Inactivity
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low bone mineral density: bone mineral density according to t and z score.
- normal bone mineral density: bone mineral density according to t and z score.

SUMMARY:
The study was conducted in the age range of 18-45 December, who were diagnosed with Cystic fibrosis.

DETAILED DESCRIPTION:
60 voluntary patients who have signed the consent form will be included. Within the scope of the research the demographic information of the individuals will be recorded. Functional capacities of individuals With the Shuttle Walking Test at Increasing Speed, respiratory functions respiratory function test, with measurements of respiratory November muscle strength and endurance, the level of dyspnea was Modified Medical Peripheral November muscle strength hand dynamometers with Research Council (mMRC) Dyspnea Scale posture assessment with the Corbin Posture Analysis Scale, trunk mobility with the Trunk Pelvis-Hip Angle Test, core stabilization with Sahrmann's Core Stability Test, individuals' perception of cosmetic deformity Walter Reed visual assessment questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-45 who were diagnosed with Cystic Fibrosis

Exclusion Criteria:

In the last year, patients;

* who had a fracture in any part of the patient's body
* who had undergone spine surgery
* who had an orthopedic, neurological or metastatic history in addition to Cystic Fibrosis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients referred by the department of chest diseases of Hacettepe University will be taken
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-01-22 (Estimated); Study Completion 2024-02-16 (Estimated)

PRIMARY OUTCOMES:
Functional Exercise Capacity | 1 day
  Functional exercise capacity by incremental shuttle walk test in patients with adult Cystic Fibrosis

SECONDARY OUTCOMES:
Posture | 1 day
  posture by Corbin Posture Analysis Form in patients with adult Cystic Fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Health Sciences Faculty, Ankara, Turkey (Türkiye)